CLINICAL TRIAL: NCT06812871
Title: A Single-arm, Multicenter, Phase 2 Study of High-dose Furmonertinib Combined With Bevacizumab and Intrathecal Pemetrexed Chemotherapy in Patients With EGFR-mutated Non-small Cell Lung Cancer and Meningeal Metastasis
Brief Title: High-dose Furmonertinib Combined With Bevacizumab and Intrathecal Pemetrexed Chemotherapy in Patients With EGFR-mutated Non-small Cell Lung Cancer and Meningeal Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li-kun Chen, Dr, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO 10120
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Non-small Cell Lung Cancer Metastatic
Keywords: EGFR mutated; meningeal metastasis
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — aflutinib; Bevacizumab; Pemetrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Furmonertinib combined with bevacizumab and intrathecal pemetrexed chemotherapy (Experimental): patients receive furmonertinib (160mg, once a day) combined with bevacizumab (7.5 mg/kg, once every 3 weeks) and pemetrexed (50 mg intrathecal injection chemotherapy, once every 3 weeks, up to 9 cycles).
  Interventions: Drug: furmonertinib

INTERVENTIONS:
Drug: furmonertinib — furmonertinib (160mg, once a day, continuous administration); bevacizumab (7.5 mg/kg body weight, once every 3 weeks); Pemetrexed (50 mg intrathecal injection chemotherapy, once every 3 weeks, up to 9 cycles).
  Other Names: bevacizumab; pemetrexed

SUMMARY:
the study conducted to evaluate the efficacy and safety of high-dose furmonertinib (160 mg qd) combined with bevacizumab and pemetrexed intrathecal chemotherapy in NSCLC patients with EGFR mutations and meningeal metastases.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological localization is NSCLC;
* confirmed EGFR exon 19 deletion mutation(19del) or EGFR exon 21L858R mutation (L858R) or EGFR exon 20 T790M mutation (T790M)）;
* Clinical diagnosis of meningeal aggravation: clinical symptoms of intracranial hypertension (headache, dizziness, vomiting, etc.) + imaging confirmation (cerebral MRI diagnosis of meningeal aggravation) or cerebrospinal fluid cytology confirmation;
* for patients with symptoms who are considered to need temporary brain local. Treatment of cough receiving adrenal corticosteroids must be kept stable or reponse for at least 1 week before the first trial of the drug preparation;
* Newly diagnosed meningeal metastasis, including meningeal metastasis after previous brain surgery and/or local radiotherapy for solid metastatic disease;
* Patients had not received previous systemic treatment for advanced NSCLC or had meningeal metastases after treatment with one third-generation EGFR-TKI.
* Obtain informed consent signed by the patient's legal representative;
* Aged ≥18 years and ≤75 years;
* Eastern Tourism Cooperation Group (ECOG) Physical condition evaluation 0-1;
* Life expectancy ≥12 week;
* Able to follow the requirements of the study protocol and confirmation procedures, and able to accept cranial wall medications;
* contraception.

Exclusion Criteria:

* Mixed non-small cell and small cell carcinoma, or squamous cell carcinoma as the main pathological type;
* Known EGFR exon 20 C797X mutation (C797X);
* history of hypersensitivity reaction to active or inactive excipients of furmonertinib, bevacizumab or pemetrexed or to drugs of similar structure or class to the investigational drug;
* Brain metastases have previously received whole-brain radiotherapy;
* Currently participating in an interventional clinical trial, or having received other study drugs or study devices within 4 weeks before the first study drug;
* Patients who have received solid organ or blood system transplantation;
* Patients with severe intracranial hypertension symptoms that cannot be relieved by discontinuation of dexamethasone and/or glycol treatment, or patients in intensive care;
* Ensure control of the patient's symptomatic pericardial, peritoneal, and pleural effusions;
* History of cancer in the last five years Other malignancies or a history of other malignancies;
* Recent active digestive events, such as duodenitis, ileitis, intestinal perforation, intestinal catheters, or other conditions that may cause gastrointestinal tract or perforation; or refractory vomiting, chronic gastrointestinal disease, inability to swallow study drugs, or previous colorectal cancer resection that prevents adequate drug absorption;
* The patient has a physique that is prone to Japanese language learning or has active Japanese language learning;Central squamous cell carcinoma orPatients at greater risk for hemoptysis; Any diamond event ≥ CTCAE grade 3, presence of open wounds, injuries or fractures in the 28th century before the first creation; if in the first Asthma was accepted 28 days before the organization meeting, the wound treatment should be evaluated by the interval period;
* History of arterial thromboembolism within the last 6 months, including vascular cerebral accident, myocardial infarction, transient cerebral contemplation;
* History of grade 4 venous thrombosis within the last 6 months, including fire embolism;
* The presence of any severe or uncontrolled systemic evidence, including difficult-to-control hypertension (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100 mmHg), uncontrolled diabetes, etc.;
* Active infections include, for example, hepatitis B, hepatitis C, and human immunodeficiency virus (HIV) infections (including those requiring intravenous therapy, active hepatitis B infection includes patients with positive hepatitis B surface test based on serological assessment and hepatitis B virus DNA >1000 copies/ml);
* previous history of interstitial lung disease, drug-induced interstitial lung disease, pneumonitis requiring steroid therapy, or any evidence of active interstitial lung disease;
* The first 28-day inspection of the drug preparation showed Lack of adequate bone marrow reserve or organ function（Within 2 weeks before blood test,No blood transfusion or blood products, granulocyte colony-stimulating factor or other hematopoietic stimulating factors were used for repair）:

  * Absolute neutrophil count <1.5 × 109/L; continuous count <100×109/L; hemoglobin <90 g/L;
  * Alanine aminotransferase > 2.5 times Upper limit of normal value (Upper limit of normal）; Aspartate aminotransferase>2.5 times ULN; Total bilirubin>1.5 times ULN;or liver transplant patients with AST and/or ALT > 5× ULN;
  * Albumin <30 g/L;
  * Serum creatinine >1.5 times ULN, and Creatinine clearance <50 mL/min（Measured or calculated by Cockcroft and Gault formula);
  * International normalized ratio (INR) > 1.5,Partially activated zymogen time（APTT>1.5 times Upper limit of normal;
  * Urine protein ≥++, and 24-hour protein >2.0g;
* Any of the following Bishop criteria:

  * Clinically significant resting electrocardiogram rhythm, respiratory, or morphological abnormalities, such as left bundle branch block, third-degree myocardial insufficiency, and second-degree myocardial insufficiency, within 28 days before the first study drug perfume;
  * Possibility Interphase Factors that increase the risk of prolonged or arrhythmic events, such as heart failure, congenital long Quantum Dots Syndrome, long Quantum Dots Family history or first-degree relatives 40 Sudden death due to coma or known prolonged Quantum Dots Any sudden or difficult to fully compensate low potassium tariffs, low tariff tariffs, and low tariff-to-tariff tariffs during the period;
  * Left ventricular ejection fraction (LVEF)Left ventricular ejection fraction）<50%, recent History of myocardial infarction, severe or unstable angina, or coronary artery bypass grafting within the past month or heart failure≥New York Heart Association (New York Heart Association (NYHA) 2 class;
* Pregnancy or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Intracranial progression-free survival | The time from receipt of study treatment to intracranial tumor PD or to death due to any cause,whichever came first, assessed up to 24 months
  The time from receipt of study treatment to intracranial tumor PD or to death due to any cause,whichever came first,

SECONDARY OUTCOMES:
systemic progression-free survival | The time from receipt of study treatment to systemic PD or to death due to any cause,whichever came first, assessed up to 24 months.
  The time from receipt of study treatment to systemic PD or to death due to any cause,whichever came first,
intracranial objective response rate | The number and percentage of objective response (PR+CR) of intracranial tumor at each time point after treatment, through study completion, an average of 12 months.
  The number and percentage of objective response (PR+CR) of intracranial tumor at each time point after treatment
overall survival | The time interval between enrollment and death from any cause,,whichever came first, assessed up to 24 months.
  The time interval between enrollment and death from any cause
safety and tolerability | adverse events will be reported and graded according to the National Cancer Institute (NCI) CTCAE version 5.0.,assessed up to 24 months.
  adverse events will be reported and graded according to the National Cancer Institute (NCI) CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No